CLINICAL TRIAL: NCT05040139
Title: A Comparative Study Between Malone Procedure and Percutaneaous Endoscopic Caecostomy in Patients Treated With Antegrade Colonic Enema for Severe Anal Incontinence and/or Constipation
Brief Title: A Comparison of Quality of Life Between MAlone Procedure and Percutaneaous Endoscopic Caecostomy in Patients With Antegrade Colonic Enema
Acronym: MAPEC
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC17_0080
Record Dates: First submitted 2018-02-26; First posted 2021-09-10 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: Constipation Aggravated; Fecal Incontinence With Fecal Urgency
Keywords: Constipation; Fecal incontinence; Antegrade colonic enema; Percutaneous Endoscopic Caecostomy; Malone Procedure
MeSH Terms: conditions — Constipation; Fecal Incontinence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Malone procedure: The percutaneous caecal access is performed surgically
  Interventions: Procedure: Malone Procedure
- Percutaneous Endoscopic Caecostomy: The percutaneous caecal acces is performed endoscopically.
  Interventions: Procedure: Percutaneous endoscopic caecostomy

INTERVENTIONS:
Procedure: Malone Procedure — Surgical procedure performed to obtain a percutaneous caecal access for the administration of antegrade colonic enemas. Briefly, the procedure is performed under general anesthesia. The surgeon bring the end of the appendix (or a tubulized segment of the ileum) out through the abdominal wall. The appendix is opened and sutured to the abdominal skin.
  Groups: Malone procedure
Procedure: Percutaneous endoscopic caecostomy — Endoscopic procedure performed to obtain a percutaneous caecal access for the administration of antegrade colonic enemas. Briefly, a coloscopy is performed to reach the caecum. The cutaneous location of the caecostomy is determined by transillumination of the caecum. A caecopexy is performed with 3 anchors at the chosen location. A specific pig-tail catheter (Chait catheter) is placed percutaneously into the caecum in the center of the 3 anchors.
  Groups: Percutaneous Endoscopic Caecostomy

SUMMARY:
Background: Antegrade colonic enema (ACE) is a second intent treatment of severe constipation and/or fecal incontinence following the failure of medical treatment. ACE is classically administered through a percutaneous access to the caecum performed surgically according to the Malone procedure (MP). Recently, a novel endoscopic approach named Percutaneous Endoscopic Caecostomy (PEC) has been proposed to perform the percutaneous access to the caecum. PEC has never been compared to the traditional MP in terms of postoperative quality of life and functional outcomes.

Objective: The aim of the study is to compare postoperative quality of life between MP and PEC in patients treated with ACE for severe constipation and/or fecal incontinence.

Hypothesis: MP and PEC achieve similar quality of life outcomes. Methods: All patients from two prospective databases who underwent MP or PEC for severe constipation and/or fecal incontinence between 2006 and 2016 will be included. They will be contacted to answer questionnaires about quality of life (GIQLI) and functional outcomes including constipation, fecal incontinence and body image assessment (KESS, Wexner and BIQ scores respectively). The main measured outcome will be GIQLI score.

Results: The results of this comparative study will determine if the endoscopic and the surgical approaches are similar in terms of quality of life, or if one of them is better than the other. This study will clarify the optimal protocol to perform a caecal percutaneous access before ACE administration in patients suffering from severe constipation and/or fecal incontinence.

DETAILED DESCRIPTION:
Background: Antegrade colonic enema (ACE) is a second intent treatment of severe constipation and/or fecal incontinence following the failure of medical treatment. ACE is classically administered through a percutaneous access to the caecum performed surgically according to the Malone procedure (MP). Recently, a novel endoscopic approach named Percutaneous Endoscopic Caecostomy (PEC) has been proposed to perform the percutaneous access to the caecum. PEC has never been compared to the traditional MP in terms of postoperative quality of life and functional outcomes.

Objective: The aim of the study is to compare postoperative quality of life between MP and PEC in patients treated with ACE for severe constipation and/or fecal incontinence.

Hypothesis: MP and PEC achieve similar quality of life outcomes. Study design: All patients from two prospective databases who underwent MP or PEC for severe constipation and/or fecal incontinence between 2006 and 2016 will be included. They will be contacted by mail to answer questionnaires about quality of life (GIQLI) and functional outcomes including constipation, fecal incontinence and body image assessment (KESS, Wexner and BIQ scores respectively). Patients who did not answer to the mail will be phoned. The collection of patients' answers will be conducted over a 3 months period.

Main outcome measures: Quality of life evaluated by the GIQLI score. Secondary outcomes measures: Functional outcomes including constipation severity (measured by the KESS score), fecal incontinence severity (measured by the Wexner score), body image impairment (measured by the BIQ score).

Results: The results of this comparative study will determine if the endoscopic and the surgical approaches are similar in terms of quality of life, or if one of them is better than the other. This study will clarify the optimal protocol to perform a caecal percutaneous access before ACE administration in patients suffering from severe constipation and/or fecal incontinence.

ELIGIBILITY:
Inclusion Criteria:

* Severe constipation and/or severe incontinence refractory to medical treatment.

Exclusion Criteria:

* Malone procedure or percutaneous endoscopic caecostomy between 2006 and 2016

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients from two prospective databases who underwent MP or PEC for severe constipation and/or fecal incontinence between 2006 and 2016 will be included. They will be contacted by mail to answer questionnaires about quality of life (GIQLI) and functional outcomes including constipation, fecal incontinence and body image assessment (KESS, Wexner and BIQ scores respectively). Patients who did not answer to the mail will be phoned. The collection of patients' answers will be conducted over a 3 months period.
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2018-11-13 (Actual); Primary Completion 2019-06-03 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Comparison of the quality of life of patients treated with anterograde colonic enemas after Malone surgical technique and percutaneous endoscopic caecostomy. | one year
  Quality of life evaluated by the GastroIntestinal Quality of Life score (GIQLI).
  The GIQLI (GastroIntestinal Quality of Life) questionnaire consists of 36 questions giving a global quality of life score and 5 sub-scores (digestive symptoms, physical scale, mental scale, social scale and effects of drug treatments).

SECONDARY OUTCOMES:
constipation | one year
  Constipation will be evaluated by the Kess constipation severity score. The Kess questionnaire consists of 11 questions assessing the symptoms of constipation and giving a single score.
anal incontinence | one year
  Anal incontinence will be evaluated with the WEXNER score.
  - The Wexner questionnaire consists of 5 questions evaluating the symptoms of incontinence and giving a single score.

CONTACTS AND LOCATIONS:
Overall Officials: Emilie Duchalais, PH, Principal Investigator — Nantes University Hospital
Locations (1):
- CHU de Nantes, Nantes, Loire-Atlantique, France